CLINICAL TRIAL: NCT04631900
Title: Effect of a Community-oriented Spiritual Intervention Programme in Persons With Depression: a Randomized Wait-list Control Trial
Brief Title: Spiritual Intervention for Persons With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City University of Hong Kong (Other)
Responsible Party: Principal Investigator, LEUNG Lai Fun Judy, Principal Investigator, City University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: judyll2222
Record Dates: First submitted 2020-11-10; First posted 2020-11-17 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Depression
Keywords: Spiritual intervention; Depression; Christian; Connectedness; randomized wait-list; community
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spiritual Intervention Programme (Experimental): The intervention is a 8 weeks' programme. The Christianity approach as the framework for spiritual intervention includes use of Bible verses, prayer, hymns singing, sharing and caring for others (mutual support) within the group.
  Through these activities, participants have opportunities to re-build and further develop their connectedness to themselves, to others, to their living, their environment, and to larger meaning and purpose.
  Interventions: Behavioral: Christianity approach as framework for spiritual intervention
- Wait-list Control group (No Intervention): Participants recruited in the waitlist control will be initially tested to generate pre-test scores and will then tested six weeks later which is equivalent to the timespan between the pre-test and post-test for the experimental spiritual programme. In between these two testing sessions, the waitlist control group will not receive any type of spiritual intervention. For ethical reasons, following the second testing session, the participants in the waitlist group will be given the opportunity to participant in the spiritual intervention programme.

INTERVENTIONS:
Behavioral: Christianity approach as framework for spiritual intervention — Intervention includes use of Bible verses, prayer, hymns singing, sharing and caring for others (mutual support) within the group. Through these activities, participants have opportunities to re-build and further develop their connectedness to themselves, to others, to their living, their environment, and to larger meaning and purpose.
  Arms: Spiritual Intervention Programme

SUMMARY:
Mental health is an integral part of health and depression has become a common and serious mental disorder. The research study aims to explore the effectiveness of spiritual intervention in persons with depression.

DETAILED DESCRIPTION:
This study aims to develop a community-oriented spiritual intervention programme that focuses on connectedness and to explore its effectiveness in persons with depression.

Objectives:

1. To evaluate the effect of this spiritual intervention on reducing depressive symptoms.
2. To evaluate the effect of spiritual intervention on enhancing hope, meaning in life, self-esteem, and social support.
3. To examine the moderatioon effect of demographic variables on the intervention effect in reducing the depressive and anxiety symptoms, and ennhancing hope, meaning in life, self-esteem, and social support.
4. To examine participant's perspectives on the healing mechanisms of the intervention.

The study is conducted as a randomized-controlled trial using a wait-list control group for comparison. The wait-list control group will receive the intervention after the completion of the post-questionnaire.

The intervention is an 8 session weekly programme. Each weekly session is around 2 hours in length and the content is as below:

1. Spirituality, mental health and depression
2. Connectedness
3. Forgiving and freedom
4. Suffering and transcendence
5. Hope
6. Gratitude
7. Relapse prevention and spiritual growth
8. Wrap-up and celebration

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese residents who can communicate in Cantonese;
* Religious or non-religious but have no objection to Christian faith rituals;
* Screening by PHQ-9 with score of 5-14 out of 27; and
* Willing to give informed consent and comply with the trial protocol.

Exclusion Criteria:

* Receiving any form of psychotherapy in the past 3 months;
* Significant cognitive impairment that is difficult to follow instructions;
* Lifetime history of psychosis that make the person unable to understand and follow instructions;
* Strong suicidal risk as rated by PHQ-9 item on suicide (score equal or more than 2), those with severe depression and strong suicidal ideas will be referred to seek professional help; and
* Adjustment of medication (antidepressant) within the past 3 months.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2021-11-27 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Change in depression measured with Patient Health Questionnaire-9 (PHQ-9) score | At baseline (T0), post at week 8 (T1) and follow-up at week 20 (T2).
  The Patient Health Questionnaire-9 (PHQ-9) (Kroenke, Spitzer, & Williams, 2001) is a self-reported questionnaire designed for use in primary care. It is a structured questionnaire that enquires after the nine symptom- based criteria for diagnostic criteria in the DSM-IV depression. Score can range from 0-27. Sum scores of 0-4 indicate none or minimal depressive symptoms, 5-9 mild depressive symptoms, 10-14 moderate depressive symptoms, and 15-27 severe depressive symptoms. It has been found to have good sensitivity and specificity (Kroenke et al., 2001). The Cronbach's alpha was reported to be 0.86 - 0.89 (Smarr & Keefer, 2011).
Change in anxiety measured with General Anxiety Disorder Questionnaire (GAD-7) | At baseline (T0), post at week 8 (T1) and follow-up at week 20 (T2).
  The General Anxiety Disorder Questionnaire (GAD-7) (Spitzer, Kroenke, Williams, & Löwe, 2006) is an easy-to-use 7 items self-administered patient questionnaire used to screen the severity measure of generalized anxiety disorder with good psychometric property. Score can range from 0-21. Sum scores of 0-5 indicates mild anxiety, 6-10 moderate anxiety, 11-15 moderately severe anxiety, and 16-21 severe anxiety. The Chinese version was tested to be a reliable and efficient instrument. (Wang Li, Lukai, Rongjing, Dayi, & Sheng, 2014).

SECONDARY OUTCOMES:
Change in hope measured with State Hope Scale (SHS) | The data will be collected in both experimental and wait-list control groups at three points: at baseline (T0), week 8 (T1) and week 20 (T2).
  The State Hope Scale (SHS) ( Snyder et al., 1996) is a 6 items self-reported instrument for measuring the extent of hope individuals held toward ongoing events in their lives. It is an 8-point Likert scale, with 1 (definitely false) to 8 (definitely true), with odd-number items measuring pathway thinking and even number items measuring agency thinking. Scores can range from 6 to 48, with higher scores representing higher hope levels.. C. R. Snyder et al. (1996) reported that SHS was a reliable and valid measure of state hope, with factor analyses confirming the two factors of agency and pathways. The internal consistency values ranging from 0.90 to 0.95 for both the agency and pathways subscale, and all adaptations and translations of the scale are reported to retain the high internal consistency (Brooks & Hirsch, 2017). The Chinese version is available (Mak, Ng, & Wong, 2011).
Change in meaning and purpose in life measured with Meaning in Life Questionnaire (MLQ) | At baseline (T0), post at week 8 (T1) and follow-up at week 20 (T2).
  The Meaning in Life Questionnaire (MLQ) (Steger, Frazier, Oishi, & Kaler, 2006) is a 10 items questionnaire. It measures 2 subscales of the presence of meaning in life and the search for meaning in life. It is a 7-point Likert scale from 1 (absolutely true) to 7 (absolutely untrue). 5 items are for presence of meaning and 5 for search for meaning. Items are summed yielding a range from 5 to 35 for each subscale with higher scores indicates a strong presence of/search for meaning in one's life. It has been translated into over two dozen languages. The Chinese version of the questionnaire has the same factor structure as the original version of MLQ among the caregivers in Hong Kong (Chan, 2014).
Change in self-esteem measured with Rosenberg Self-Esteem Scale (RSES) | At baseline (T0), post at week 6 (T1) and follow-up at week 18 (T2).
  The Rosenberg Self-Esteem Scale (RSES) (Rosenberg, 1965) is a widely used instrument (10 items) around the world for measuring self-esteem with a 4 point Likert scale ranging from ranging from 4 (strong agree) to 1 (strong disagree). Reverse scoring (4= strongly disagree to 1= strongly agree are used for five negatively worded items: 2, 5, 6, 8 and 9. The total score ranges from 10 to 40 with higher scores indicates higher self-esteem. The internal reliability and factor structure of the scale is psychometrically sound across many languages and cultures (Schmitt & Allik, 2005).
Change in perceived social support measured with Multidimensional Scale of Perceived Social Support (MSPSS) | At baseline (T0), post at week 8 (T1) and follow-up at week 20 (T2).
  The Multidimensional Scale of Perceived Social Support (MSPSS) (Zimet, Dahlem, Zimet, & Farley, 1988) is one of the most extensively used instruments to assess social support. It is a 12 items self -administered measure of social support with 3 subscales of family, friends, and significant others. It is a 7 point Likert scale ranging from 1(very strongly disagree ) to 7 (very strongly agree). The mean scores for significant other subscale is the sum across items 1, 2, 5 & 10, then divided by 4; the mean scores for family subscale is the sum across items 3,4, 8, & 11, then divided by 4; the mean scores of friends subscale is the sum across items 6, 7, 9, &b 12, then divided by 4. The mean score of the total scale is the sum across all 12 items, then divided by 12. The mean score range from 1 (lowest) to 7 (highest). The Chinese version of MSPSS has good internal consistency reliability with composite reliability values of more than 0.7 (Y. Wang, Wan, Huang, Huang, & Kong, 2017).

OTHER OUTCOMES:
Change in spiritual experience measured with Daily Spiritual Experience Scale (DSES) | At baseline (T0), post at week 8 (T1) and follow-up at week 20 (T2).
  The Daily Spiritual Experience Scale (DSES) (Underwood, 2011) is a 16-items self-reported validated questionnaire that assesses ordinary experience of the transcendence in daily life. It includes constructs such as awe, gratitude, mercy, sense of connection with the transcendent and compassionate love. It also includes measures of awareness of inspiration and a sense of deep inner peace. The first 15 items are scored with a Likert scale, from many times a day for 6 marks to never or almost never for 1 mark. The last item has only four response ranging from as close as possible for 4 mark to not close for 1 mark. The scores are summed up with higher score indicate higher level of spirituality. The reliability and validity of DSES have been tested to be satisfactory (Underwood & Teresi, 2002). It has been translated into over 40 languages. The Chinese version of DSES has been found to have the satisfactory psychometric properties (Ng, Fong, Tsui, Au-Yeung, & Law, 2009).

CONTACTS AND LOCATIONS:
Overall Officials: Judy LF LEUNG, PhD(c), Principal Investigator — City University of Hong Kong
Locations (1):
- City University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) from completed clinical trials should be responsibly shared to support efficient clinical research, generate new knowledge and bring benefit to patients. The result can be disseminated via seminars, conference presentations, and various media.
Supporting Information: Study Protocol, SAP
Time Frame: The completion of the data collection should be finished by Dec 2021 and time frame of sharing individual participant data (IPD) should be by Dec 2022.
Access Criteria: It is hoped that the result can be disseminated via seminars, conference presentations and various media. The actual website is not available at the moment.

REFERENCES:
- [Background] Chan WC. Factor structure of the Chinese version of the Meaning in Life Questionnaire among Hong Kong Chinese caregivers. Health Soc Work. 2014 Aug;39(3):135-43. doi: 10.1093/hsw/hlu025. PMID 25095626
- [Background] Brooks, B. D., & Hirsch, J. K. (2017). State Hope Scale. In V. Zeigler-Hill & T. K. Shackelford (Eds.), Encyclopedia of Personality and Individual Differences (pp. 1-4). TN: Springer International Publishing.
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Li, W., Lukai, Rongjing, D., Dayi, H., & Sheng, L. (2014). GW25-e4488 The value of Chinese version GAD-7 and PHQ-9 to screen anxiety and depression in cardiovascular outpatients. JACC (Journal of the American College of Cardiology), 64(16), C222-C222. doi:10.1016/j.jacc.2014.06.1038
- [Background] Mak WW, Ng IS, Wong CC. Resilience: enhancing well-being through the positive cognitive triad. J Couns Psychol. 2011 Oct;58(4):610-7. doi: 10.1037/a0025195. PMID 21895357
- [Background] Rosenberg, M. (1965). Society and the adolescent self-image. Princeton, N.J.: Princeton University Press.
- [Background] Schmitt DP, Allik J. Simultaneous administration of the Rosenberg Self-Esteem Scale in 53 nations: exploring the universal and culture-specific features of global self-esteem. J Pers Soc Psychol. 2005 Oct;89(4):623-42. doi: 10.1037/0022-3514.89.4.623. PMID 16287423
- [Background] Smarr KL, Keefer AL. Measures of depression and depressive symptoms: Beck Depression Inventory-II (BDI-II), Center for Epidemiologic Studies Depression Scale (CES-D), Geriatric Depression Scale (GDS), Hospital Anxiety and Depression Scale (HADS), and Patient Health Questionnaire-9 (PHQ-9). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S454-66. doi: 10.1002/acr.20556. No abstract available. PMID 22588766
- [Background] Snyder CR, Sympson SC, Ybasco FC, Borders TF, Babyak MA, Higgins RL. Development and validation of the State Hope Scale. J Pers Soc Psychol. 1996 Feb;70(2):321-35. doi: 10.1037//0022-3514.70.2.321. PMID 8636885
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Steger, M. F., Frazier, P., Oishi, S., & Kaler, M. (2006). The Meaning in Life Questionnaire: Assessing the Presence of and Search for Meaning in Life. Journal of Counseling Psychology, 53(1), 80-93. doi:10.1037/0022-0167.53.1.80
- [Background] Wang Y, Wan Q, Huang Z, Huang L, Kong F. Psychometric Properties of Multi-Dimensional Scale of Perceived Social Support in Chinese Parents of Children with Cerebral Palsy. Front Psychol. 2017 Nov 21;8:2020. doi: 10.3389/fpsyg.2017.02020. eCollection 2017. PMID 29209254
- [Background] Zimet, G. D., Dahlem, N. W., Zimet, S. G., & Farley, G. K. (1988). The Multidimensional Scale of Perceived Social Support. Journal of Personality Assessment, 52(1), 30-41. doi:10.1207/s15327752jpa5201_2Zimet, G. D., Dahlem, N. W., Zimet, S. G., & Farley, G. K. (1988). The Multidimensional Scale of Perceived Social Support. Journal of Personality Assessment, 52(1), 30-41. doi:10.1207/s15327752jpa5201_2